CLINICAL TRIAL: NCT00083252
Title: Study of Talabostat and Cisplatin in Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Point Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTH-303
Record Dates: First submitted 2004-05-14; First posted 2004-05-18 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Melanoma; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — talabostat; Tablets; Cisplatin

INTERVENTIONS:
Drug: talabostat (PT-100) tablets
Drug: cisplatin

SUMMARY:
The purpose of this study is to assess the antitumor activity and safety of the combination of talabostat and cisplatin in patients with metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma that is metastatic (unresectable Stage IV per AJCC 2002)
* Patients with measurable disease defined as at least one measurable index lesion with clearly defined margins
* ECOG Performance Status of 0, 1, or 2
* Expected survival ≥12 weeks
* Written informed consent

Exclusion Criteria:

* More than 1 prior chemotherapy or biotherapy regimen for metastatic melanoma
* Radiation therapy to >50% of the bone marrow. Patients must not have had prior radiotherapy to index lesions unless they have clearly progressive disease in this site or there is measurable disease outside the area of prior radiation.
* Clinically significant laboratory abnormalities
* Symptomatic CNS metastases
* Any malignancy within the 5 years immediately prior to the first dose of study medication with the exception of basal cell or non-metastatic squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix
* The need for chronic (i.e., >7 days) oral or intravenous corticosteroid therapy
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol
* Patients who are within 30 days of chemotherapy, radiation therapy, immunotherapy, or other investigational medication for melanoma. Patients must have recovered from all of the side effects of treatment in order to be enrolled.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Cancer Institute Medical Group, Inc., Santa Monica, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Cancer Center of Florida, Ocoee, Florida
  - Indiana Hematology Oncology Consultants, Indianapolis, Indiana
  - New Mexico Cancer Center Alliance, Albuquerque, New Mexico
  - NYU School of Medicine, New York, New York
  - Fifth Avenue Medical Healthcare, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Cancer Care Northwest Research, Spokane, Washington